CLINICAL TRIAL: NCT06058182
Title: RNA as Prognostic Biomarkers in Patients With Acute Coronary Syndrome
Acronym: RNAacs
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Luca Testa, Principal investigator, IRCCS Policlinico S. Donato
Other Study IDs: RNA_ACS
Record Dates: First submitted 2023-02-15; First posted 2023-09-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood draws — Pre-procedure, post-procedure (12-24 h), 6-month, and 12-month blood draws

SUMMARY:
Identify circulating protein-coding (mRNAs) or non-coding (ncRNAs) transcripts (ACS_signature) predictive of ventricular dysfunction in ACS patients undergoing PCI.

DETAILED DESCRIPTION:
Perform an observational, prospective study involving the evaluation of circulating biomarkers predictive of ventricular dysfunction (FE <45%) in patients with ACS.

In particular, will be to verify whether there are circulating transcripts in peripheral blood, coding or not for proteins (mRNAs or ncRNAs), modulated differently in patients with ACS (ACS_signature) undergoing PCI, distinguished on the basis of evolution towards ventricular dysfunction. The study will be based on whole genome transcriptomic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients with ACS (first episode), defined according to the guidelines of the European Society of Cardiology (ESC) 2017
3. Indication for percutaneous revascularization treatment
4. Informed consent to study enrollment

Exclusion Criteria:

1. Severe valve disease or other conditions requiring cardiac surgery
2. Previous cardiac surgery including coronary artery bypass grafts
3. Total chronic occlusions
4. Patients with known hypersensitivity or contraindication to any of the following drugs:

   * heparin
   * aspirin,
   * clopidogrel,
   * ticlopidine,
   * sirolimus,
   * everolimus.
5. Any contraindication to drug-eluting stent implantation (DES)
6. Patients with a documented history of myocardial infarction;
7. Left ventricular ejection fraction (LVEF) <30% before PCI
8. Patients in cardiogenic shock
9. Patients with advanced ST-segment elevation myocardial infarction (> 48 h from onset of symptoms/Q waves on electrocardiogram) or undergoing fibrinolysis;
10. Patients with prior known cardiomyopathy with LVEF < 40%
11. Patients with malignant neoplasm or systemic disease with quoad vitam prognosis less than 1 year;
12. Patients with known active infectious diseases;
13. Patients who are unable to express valid informed consent to the act of enlistment
14. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study, observational, prospective, single center that will make use of the recruitment of consecutive patients with acute coronary syndrome treated with angioplasty
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
identify circulating transcripts codifying and not for mRNA proteins, predictive of ventricular dysfunction in patients with acute coronary artery syndrome treated with coronary angioplasty. | 1 years
  For discovery activities using RNA-sequencing, based on literature data, we assume a sample size of 40 patients (20 per group) that will allow to evaluate the 40 transcripts that differentiate patients with ventricular dysfunction and not ventricular dysfunction, out of a total of 17,500 tests, with a power of 94.0 %, an FDR value of 0.02. For qPCR validation activities, a power of 95% is obtained by analyzing 50 samples per group by evaluating differences between the averages of 2,2 times, with α= 0,01 and σ= 1,4.

SECONDARY OUTCOMES:
Evaluate the association of the ACS_signature with possible adverse events at 12 months and its prognostic ability in the prediction of adverse events additional to the use of standard clinical parameters. | 1 years
  Adverse events are defined: death from cardiovascular causes, re infarction, non-fatal stroke, new coronary revascularization, arrhythmias, development of heart failure and new hospitalizations for cardiovascular causes

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico S. Donato, Milan, Italy, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-01-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT06058182/Prot_000.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT06058182/ICF_001.pdf